CLINICAL TRIAL: NCT01990040
Title: A Prospective, Multi-center Registry for Patients With Short Bowel Syndrome
Brief Title: Registry for Participants With Short Bowel Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: TED-R13-002; EUPAS7973 (Other: ENCePP EU PAS)
Record Dates: First submitted 2013-11-11; First posted 2013-11-21 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; SBS; teduglutide; Gattex
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Teduglutide treated: SBS participants who have been treated with teduglutide.
- Non-teduglutide treated: SBS participants who have not been treated with teduglutide.

SUMMARY:
This is a global prospective, observational, multi-center registry to evaluate the long-term safety profile for participants with short bowel syndrome (SBS) who are treated with teduglutide in a routine clinical setting. The registry will also evaluate the long-term clinical outcomes in participants with SBS. SBS participants treated and not treated with teduglutide will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, of any age, with a diagnosis of short bowel syndrome (SBS).
2. Signed informed consent and medical records release by the participant or a legally acceptable representative
3. Participants who have never received teduglutide treatment must be on parenteral nutrition (PN)/intravenous (IV) fluids support for at least 6 months at the time of enrollment.

Exclusion criteria:

1. Participants currently participating in a blinded clinical trial or their extension studies.
2. Participants who have never been on PN/IV support.
3. Participants who are currently or previously exposed to any Glucagon-like peptide 2 (GLP-2) analogs other than teduglutide.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This registry is to enroll both male and female adult participants, of any age, with a diagnosis of SBS.
Sampling Method: Non-Probability Sample
Enrollment: 1806 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Colorectal Cancer in Short Bowel Syndrome (SBS) Participants With a Remnant Colon Currently Being Treated With or Ever Having Been Treated With Teduglutide | 10 years
  Incidence rates of colorectal cancer in participants will be calculated by dividing the number of incident colorectal cancer cases by the total number of person-years observed since beginning treatment with teduglutide.

SECONDARY OUTCOMES:
Occurrence of Other Malignancy | 10 years
  Incidence rates of other malignancies will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Benign Neoplasia of the Gastrointestinal (GI) tract, Hepatobiliary System, and Pancreas in Participants | 10 years
  Incidence rates of benign neoplasia of the GI tract, hepatobiliary system, and pancreas will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Colorectal Polyps | 10 years
  Incidence rates of colorectal polyps will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Intestinal Obstruction | 10 years
  Incidence rates of intestinal obstruction will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Pancreatic and Biliary Disease | 10 years
  Incidence rates of pancreatic and biliary disease will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Heart Failure and Other Manifestations of Volume Overload | 10 years
  Incidence rates of heart failure and other manifestations of volume overload will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Allergic/Hypersensitivity Reaction to Teduglutide | 10 years
  Incidence rates of allergic/hypersensitivity reactions to teduglutide will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide.
Occurrence of Other Adverse Events (AEs) Potentially Related to Treatment with Teduglutide | 10 years
  Incidence rates of other AEs will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide. Incidence rates of other AEs will be calculated by dividing the number of incident cases by the total number of person-years observed since beginning treatment with teduglutide. An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product (ICH Guidance E2A 1995). This includes an exacerbation of a pre-existing condition.
Actual Volume Change in Parenteral Support (PS) | 10 years
  PS will be measured by parenteral treatment volume (liters/week) and days (days/week) that occurred in the 7 days prior to the visit.
Percentage Volume Change in Parenteral Support (PS) | 10 years
  PS will be measured by parenteral treatment volume (liters/week) and days (days/week) that occurred in the 7 days prior to the visit.
Actual Change in the Number of Days per Week on Parenteral Support (PS) | 10 years
  PS will be measured by parenteral treatment volume (liters/week) and days (days/week) that occurred in the 7 days prior to the visit.
Percentage Change in the Number of Days per Week on Parenteral Support (PS) | 10 years
  PS will be measured by parenteral treatment volume (liters/week) and days (days/week) that occurred in the 7 days prior to the visit.
Percent of Participants Weaning From Parental Support (PS) | 10 years
  PS will be measured by parenteral treatment volume (liters/week) and days (days/week) that occurred in the 7 days prior to the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Shire, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b600e4db2bf003ab48d50